CLINICAL TRIAL: NCT04670757
Title: One Centre, Single Ascending Dose and Double Blind Multiple Ascending Dose, Safety and Pharmacokinetics Phase I Study of CPL409116 Compound in Healthy Volunteers.
Brief Title: Safety and Pharmacokinetics of JAK/ROCK Inhibitor in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celon Pharma SA (Industry)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 01JAK2020
Record Dates: First submitted 2020-11-27; First posted 2020-12-17 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-04

CONDITIONS: Healthy
Keywords: Pharmacokinetics; JAK inhibitors; ROCK inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Only Phase IB is to be double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPL409116 (Experimental): PART A. IMP is to be administered orally in single ascending dose in the groups consisting of 3 volunteers according to '3+3' design'. Dose escalation scheme is to be determined based on preclinical results and due to dose limiting observation (DLT).
  PART A additional. Assessing the effect of food on bioavailability of CPL409116. IMP is to be administered orally in single dose in fasted and fed state in the group of 12 volunteers.There is to be one week wash-out between two treatment periods for this cohort.
  Interventions: Drug: CPL409116
- PLACEBO (Experimental): PART B. Two participants from each of 4 cohorts (total of 8 participants) are to receive masking placebo tablet once daily for 14 days. There is to be dose escalation between cohorts. Participants are to be randomized within cohorts.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CPL409116 — IMP administration, tablets contain CPL409116 as an active ingredient
  Arms: CPL409116
Drug: Placebo — Placebo comparator
  Arms: PLACEBO

SUMMARY:
The aim of the following clinical trial is to determine safety an pharmacokinetic parameters in healthy volunteers after oral administration of Janus kinases and Rho-kinases inhibitor (JAK/ROCKi), called CPL409116.Janus kinase (JAK) inhibitors are a new class of small molecule drugs that modulate inflammatory pathways by blocking one or more JAK receptors. In recent years, JAK inhibitors have emerged as a new option for the treatment of various inflammatory diseases, including rheumatoid arthritis, psoriatic arthritis, spondyloarthritis, skin disorders and others. CPL409116 inhibits JAK1 and JAK3 with less inhibitory activity against JAK2 and Tyk2. Inhibition of these kinases decreases inflammatory cytokine release which in turn decreases lymphocyte activation and proliferation. Moreover, CPL409116 blocks Rho-kinases (ROCKs), which are involved in diverse cellular processes including actin cytoskeleton organization, cell adhesion and motility, proliferation, apoptosis as well as smooth muscle contraction. ROCKs signalling is one of the major pathways implicated in the pathogenesis of cardiovascular, renal as well as fibrotic diseases. However recent data indicate their role in immune cell regulation and inflammatory disease development. CPL409116 was designed predominantly for the therapy of immune-related diseases: rheumatoid arthritis, psoriasis and because antifibrotic therapies are needed. Dual inhibition of JAK/ROCK kinases may be beneficial for patients suffering from fibrotic complications of inflammatory disease.

Rheumatoid arthritis (RA) is a chronic systemic autoimmune disease characterised by persistent joint inflammation leading to loss of joint function as well as cartilage and bone damage. Chronic, progressive course of the disease results in disability, reduced quality of life, as well as higher comorbidity and mortality rates. It is well documented that JAK kinases play a pivotal role in cytokine receptor signalling to phosphorylate and activate signal transducer and activator of transcription (STAT) proteins. Several of these JAK-controlled cytokine receptor pathways are immediately involved in the initiation and progression of RA pathogenesis. Cytokines promote autoimmunity, maintain chronic inflammatory synovitis and drive the destruction of joint tissue. In consequence on the basis of the preclinical study results the IMP with the active ingredient CPL409116 has been classified as a good clinical candidate for the treatment of RA.

DETAILED DESCRIPTION:
The following clinical trial consists of two phases IA and IB. Approximately 68 volunteers who meet all the inclusion and none of the exclusion criteria are going to be enrolled into the study. Phase IA (approx. 24 male and female volunteers) is to evaluate safety and tolerability after single oral administration of the Investigational Medicinal Produkt (IMP) to healthy volunteers. Additional cohort (approx 12 healthy volunteers) is going to be included in the phase IA of the study to assess the food effect on CPL409116 compound's bioavailability after one dose of single oral IMP administration. There are to be two treatments periods for this cohort: fasted and fed. Phase IB (approx. 32 male and female volunteers) is to evaluate safety and tolerability after two weeks of oral administration of IMP to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Body-mass index (BMI): ≥ 18.5 kg/m² and < 29.9 kg/m²,
2. Physical examination (such as observation, palpation, percussion and auscultation) without any clinically relevant abnormality,
3. Clinical laboratory results in hematology or renal/hepatic test and clinical laboratory results in other tests without any clinically relevant abnormalities as assessed by Investigator,
4. Non-smoker and non-user of tobacco products for at least 3 months before screening,
5. Subject able to provide written informed consent after receiving information about the trial,
6. Informed Consent Form signed and dated prior to Screening evaluations,
7. Ability and willingness to comply with the requirements of the study protocol,
8. Volunteer (or his/her partner) of childbearing potential willingness to use acceptable forms of contraception: complete abstinence from sexual intercourses or barrier method of spermicide (condom, diaphragm) or intrauterine device or hormonal contraceptive since at least screening evaluations for male volunteers and since at least 4 weeks before screening for female volunteers. Volunteers are furthermore willing to use it for 90 days (males) or 30 days (females) after examination at the end of the study.
9. Negative result of the COVID-19 RT-PCR test (real-time reverse transcription polymerase chain reaction) for the qualitative detection of nucleic acid from SARS- CoV-2 before inclusion to the study.

Exclusion Criteria:

1. Subject with known allergy, hypersensitivity, intolerance or contraindication to other drugs similar in structure or class to CPL409116 compound, or to any excipients of the formulation,
2. Any known significant current or past acute or chronic disease or condition of the: circulatory, respiratory, hematopoietic, endocrine, nervous and musculoskeletal system, alimentary and urinary tracts, allergic disease, genetic or psychiatric disorder, thromboembolism in a volunteer or in members of their close family that could influence the present general health condition, at the Investigator's discretion,
3. Thrombophilia or genetic predisposition to thrombophilia in a volunteer and/or previous or current thromboembolic events/ disease in a volunteer or in members of their family,
4. Subject has a long QT interval analysis syndrome or is under the treatment with antiarrhythmic drugs,
5. Current disease of the alimentary tract, liver or kidneys that may influence absorption, distribution and/or elimination of the studied drug, as assessed by the Investigator and documented in the medical history,
6. Medical condition that requires administration of other drugs or use of any drug within the 4 weeks preceding the first IMP administration and during the entire study. Drugs commonly used with fast metabolism may be administered and is up to Investigator discretion (i.e. pain killers),
7. Participation in other clinical trials, where at least one dose of study drug was administered, within 90 days preceding the screening phase,
8. Blood drawn within 30 days prior to inclusion in this study (more or equal to 300 mL),
9. Positive results from pregnancy test in female volunteers,
10. Lactation in female volunteers,
11. Hypotension or hypertension in medical history, on Screening Day or before treatment period, if Principal Investigator is to assess it as clinically relevant,
12. Narcotic and alcohol addiction or abuse (more than 14 alcohol units per week: one unit = 150 mL wine, 360 mL beer, 45 mL 40 % spirits) (UK guidelines),
13. Positive results of HBsAg, anti-HCV or anti-HIV tests,
14. Positive drug screen or alcohol breath tests,
15. Subjects who adhere to a special diet (e.g. low calories, vegetarian, etc.),
16. The subject is considered by the Investigator to be an unsuitable candidate to participate in the study for any reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Determination of maximum tolerated dose (MTD) or administration of the maximum dose provided in the protocol after single and multiple oral administration of IMP. | up to 48 hours after single administration of IMP in PART A and up to 48 hours after the last IMP administration in PART B
  MTD is defined as the highest dose for which no more than 1 of the 6 treated volunteers (less than 1/3) exhibits dose limiting toxicity (DLT).
Safety and tolerability of IMP after single and multiple oral administration | up to 14 days in Part A and after multiple oral IMP administration up to 28 days in Part B
  Participants during hospitalization are to be closely observed to assure maximal safety and to collect occurrence of all adverse event. To follow-up on all study participants telephone calls with a request for information regarding their health condition are to be made.

SECONDARY OUTCOMES:
Cmax - maximum plasma concentration | up to 48 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 8 in PART B and up to 48 hours after the last IMP administration on Day 14 in PART B]
  The maximum concentration of the CPL409116 compound in plasma after IMP administration, obtained directly from the measured concentrations.
AUC(0-48) - area under the plasma concentration - time curve from time 0 to 48h after IMP administration | up to 48 hours after administration of IMP in PART A
  The AUC(0-48) is a measure of total plasma exposure to the drug from time point zero to 48 hours after IMP administration
AUC(0-24) - area under the plasma concentration - time curve from time 0 to 24h after IMP administration | up to 24 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1 and 8 in PART B
  The AUC(0-24) is a measure of total plasma exposure to the drug from time point zero to 24 hours after IMP
AUC(0-inf) - area under the plasma concentration - time curve from time 0 to infinity time | up to 48 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 8 in PART B and up to 48 hours after the last IMP administration on Day 14 in PART B
  The AUC(0-inf) is a measure of total plasma exposure to the drug from time point zero extrapolated to infinity.
Tmax - time to reach maximum concentration | 48 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 8 in PART B and up to 48 hours after the last IMP administration on Day 14 in PART B
  The Tmax is time to reach the maximum plasma concentration (Cmax), obtained directly from the actual sampling times.
Kel - terminal elimination rate constant | up to 48 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 8 in PART B and up to 48 hours after the last IMP administration on Day 14 in PART B
  Kel is to be estimated via linear regression of time versus log of concentration
T1/2 - The plasma elimination half-life | up to 48 hours after administration of IMP in PART A and up to 24 hours after the IMP administration determined on Day 1, 8 in PART B and up to 48 hours after the last IMP administration on Day 14 in PART B
  T1/2 is to be calculated as 0.693/Kel.
C (1,t) - CPL409116 concentration | Determined on Day 2, 3, 4, 5, 6, 7, 9, 10, 11, 12 and 13 in Part B
  The concentration of CPL409116 on day t before product administration.
C (Tmax, t) - CPL409116 concentration | Determined on Day 2, 3, 4, 5, 6, 7, 9, 10, 11, 12 and 13 in Part B
  The concentration on day t measured on time Tmax which was calculated in PART A of the study

CONTACTS AND LOCATIONS:
Locations (1):
- BioResearch Group Sp. z o.o., Kajetany, Nadarzyn, Poland

REFERENCES:
- [Derived] Rudzki PJ, Jarus-Dziedzic K, Wlodarczyk D, Kaza M, Pankiewicz P, Gierczak-Pachulska A, Banach M, Zygmunt B, Piwowarczyk C, Zero P, Rabczenko D, Segiet-Swiecicka A, Wieczorek M. First-in-human study of CPL'116 - a dual JAK/ROCK inhibitor - in healthy subjects. Front Pharmacol. 2025 Apr 1;16:1583723. doi: 10.3389/fphar.2025.1583723. eCollection 2025. PMID 40235539
- See also: The rationale for Janus kinase inhibitors for the treatment of spondyloarthritis — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC6343466/